CLINICAL TRIAL: NCT05930353
Title: Psychometric Validation of a French-language Version of the PERMA-Profiler: Tools for Assessing Multidimensional Subjective Well-being
Acronym: PERMAPROFILER2
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2023/JJ-01
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: COHORT — this evaluation includes a brief interview with perma profiler scale

SUMMARY:
The main objective of this study is to carry out the psychometric validation of the PERMA-Profiler in a population representative of the general French population and in comparison with the reference questionnaire The PERMA-Profiler.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years).
* Person able to read and understand French
* Person willing to participate in this study

Exclusion Criteria:

* The person does not understand the French language
* Person has a history of traumatic brain injury
* The person refuses to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general population
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PERMA PROFILER French Version: diagnostic properties | DAY 0
  sensitivity, specificity

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No